CLINICAL TRIAL: NCT04597125
Title: A Phase 4, Randomized, Open-label, Multicenter Efficacy and Safety Study of Standard Dose of Radium-223 Dichloride vs. Standard Doses of Novel Anti-hormonal Therapy (NAH) in Patients With Bone Dominant Metastatic Castration Resistant Prostate Cancer (mCRPC) Progressing on/After One Line of NAH
Brief Title: RADIANT: A Study of Radium-223 Dichloride (Xofigo) vs Enzalutamide or Abiraterone (ARPIs, Androgen Receptor Pathway Inhibitors) in Patients With Prostate Cancer That Has Spread to the Bones (mCRPC, Metastatic Castration-Resistant Prostate Cancer)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20510; 2023-505830-89-00 (Other: CTIS (EU)); 2019-000476-42 (EudraCT Number)
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castrate Resistant Prostate Cancer (mCRPC)
MeSH Terms: interventions — radium Ra 223 dichloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Participants with bone dominant metastatic castration resistant prostate cancer (mCRPC) progressing on/after one line of NAH will be randomized to receive radium-223 dichloride
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)
- Arm B (Active Comparator): Participants with bone dominant metastatic castration resistant prostate cancer (mCRPC) progressing on/after one line of NAH will be randomized to receive second novel anti-hormonal therapy (NAH)
  Interventions: Drug: NAH therapy

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Participants will receive Radium-223 (BAY88-8223) every 4 weeks for a total of 6 administrations via intravenous (IV) injection
  Arms: Arm A
Drug: NAH therapy — Participants will receive continuous NAH (either Abiraterone acetate plus prednisone/prednisolone [AAP] or enzalutamide) by mouth (per os) daily
  Other Names: Second novel anti-hormonal therapy
  Arms: Arm B

SUMMARY:
Researchers in this study want to compare how well drug radium-223 dichloride (Xofigo) and new (novel) anti-hormonal (NAH) therapy work in participants with prostate gland cancer which has spread to the bone and progressed on or after one line of NAH therapy. Meanwhile researchers want to compare the safety of radium-223 dichloride and NAH therapy. Radium-223 dichloride is known as a radioactive drug that is taken up by bones after it is injected into the body. It works by giving off a type of radioactivity that travels a very short distance and kills the tumor cells that have spread to the bone without major effects to the healthy cells. It has been approved in many countries for the treatment of patients with prostate cancer which has spread to the bone. The NAH drugs used in this study will be either abiraterone acetate (Zytiga) (plus prednisone/prednisolone) or enzalutamide (Xtandi). Both of them are standard approved medications which are used in the treatment of advanced prostate cancer.

Participants in this study will receive either Radium-223 dichloride or a NAH therapy. Radium-223 dichloride will be given as an infusion into one of the veins on Day 1 of each 4-week cycle for a total of up to 6 cycles. Oral NAH therapy will be given per the standard approved dose once daily until the disease has progressed. Participants will visit the hospital or clinic every 2 weeks for the first 6 cycles, and only on the first day of each cycle from cycle 7 and onwards. Observation for each participant will last for about 2 years in total. Blood and urine samples will be collected from the participants and participants will be asked to complete questionnaires about the well-being and the pain.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have histologically confirmed adenocarcinoma of the prostate.
* Participants with mCRPC progressing on/after one line of an approved NAH (eg. abiraterone, enzalutamide, apalutamide, or darolutamide, after being treated for at least 3 months) in an authorized prostate cancer indication.
* One prior taxane treatment regimen (at least 2 cycles) for metastatic prostate cancer (mHSPC and mCRPC) or refusal or ineligibility of such a regimen.
* Prostate cancer progression documented by PSA according to the Prostate Cancer Working Group 3 (PCWG3) criteria or radiological progression according to RECIST, version 1.1.
* At least 2 bone metastases on bone scan within 4 weeks prior to randomization with no current or history of lung, liver, other visceral, and / or brain metastasis.
* Symptomatic prostate cancer. A worst pain score (WPS) of at least 1 on the Brief Pain Inventory-Short Form (BPI-SF) Question #3 (worst pain in last 24 hours). This is to be assessed once during the Screening period.
* Maintenance of medical castration or surgical castration with testosterone less than 50 ng/dL (1.7 nmol/L). If the participant is being treated with luteinizing hormone releasing hormone (LHRH) agonists or antagonists (participant who has not undergone orchiectomy), this therapy must have been initiated at least 4 weeks prior to randomization and must be continued throughout the study.
* Participants must be on a BHA treatment, such as bisphosphonates or denosumab treatment unless such treatment is contraindicated or not recommended per investigator's judgement and inclusion is agreed to by the medical monitor.
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1.
* Life expectancy ≥ 6 months.
* Able to swallow abiraterone and prednisone/prednisolone or enzalutamide as whole tablets/capsules.
* Laboratory requirements:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
  * Platelet count ≥ 100 x 10^9/L
  * Hemoglobin (Hb) ≥ 9.0 g/dL (90 g/L; 5.6 mmol/L)
  * Total bilirubin level ≤ 1.5 x institutional upper limit of normal (ULN) (except for participants with documented Gilbert's disease)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
  * Creatinine ≤ 1.5 x ULN or estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m^2 as calculated using the Cockcroft-Gault equation
  * International normalized ratio (INR) of prothrombin time (PT; PT-INR) and partial thromboplastin time (PTT) ≤ 1.5 times the ULN. Participants treated with warfarin or heparin will be allowed to participate in the study if no underlying abnormality in coagulation parameters exists per prior history; weekly evaluation of PT-INR / PTT will be required until stability is achieved (as defined by local standard of care and based on pre-study PT-INR / PTT values)
  * Serum albumin > 30 g/L
  * Serum potassium ≥ 3.5 mmol/L
* Capable of giving signed informed consent

Exclusion Criteria:

* Active infection or other medical condition that would make prednisone / prednisolone (corticosteroid) use contraindicated.
* Any chronic medical condition requiring a higher dose of corticosteroid than 10 mg prednisone / prednisolone equivalent daily for more than 2 months.
* Pathological finding consistent with tumors with predominant neuroendocrine features or small cell carcinoma of the prostate.
* History of osteoporotic fracture
* History of visceral metastasis, or presence of visceral metastasis detected by screening imaging examinations.
* History of or known brain metastasis.
* Malignant lymphadenopathy exceeding 3 cm in short-axis diameter.
* Other malignancy treated within the last 3 years (except non-melanoma skin cancer or low-grade superficial bladder cancer)
* Imminent spinal cord compression based on clinical findings and / or magnetic resonance imaging (MRI). Participants with history of spinal cord compression should have completely recovered.
* Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 95 mmHg). Participants with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment.
* Active or symptomatic viral hepatitis
* History of pituitary or adrenal dysfunction
* Any other serious illness or medical condition such as, but not limited to:

  * Any infection ≥ National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 Grade 2
  * Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class II to IV heart disease or cardiac ejection fraction measurement of <50% at baseline
  * Current clinical evidence of any uncontrolled cardiac arrhythmia
  * Crohn's disease or ulcerative colitis
  * Bone marrow dysplasia
  * Moderate and severe hepatic impairment (Child-Pugh Classes B and C)
  * Unmanageable fecal incontinence.
* Any condition, which in the opinion of the investigator would preclude participation in this trial (eg, history of seizure).
* Hypersensitivity to the active substances or to any excipients of radium-223 dichloride, or abiraterone acetate or enzalutamide.
* Prior therapeutic systemic radiation with any radiopharmaceutical medication for the treatment of prostate cancer, including but not limited to lutetium-177, strontium-89, samarium-153, iodine-131, rhenium-186, rhenium-188, or radium-223. Radiopharmaceutical compounds used for diagnosis purposes only are allowed.
* Prior hemibody external radiotherapy is excluded. Participants who received other types of prior external radiotherapy are allowed provided that the bone marrow function is assessed and meets the protocol requirements for Hb, ANC, and platelet count.
* Blood transfusion or erythropoietin stimulating agents 4 weeks prior to Screening and during the whole Screening period before randomization.
* Excessive intake of biotin above the recommended daily dose of 30 μg. Biotin is found in multivitamins, including prenatal multivitamins, biotin supplements, and dietary supplements for hair, skin, and nail growth at levels that may interfere with laboratory tests.
* Prior administration of an investigational therapeutic for CRPC.
* Previous (within the last 4 weeks of randomization) or concurrent participation in any interventional clinical study with investigational study drug administration.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to five years

SECONDARY OUTCOMES:
Time to first symptomatic skeletal event (SSE) | Up to five years
Radiological Progression-free survival (rPFS) | Up to five years
  rPFS is defined as the time from the date of randomization to the date of confirmed radiological progression or death, whichever occurs first.
Time to pain progression (BPI-SF) | Up to five years
  The Brief Pain Inventory-Short Form (BPI-SF) is a self-administered questionnaire with 11 items designed to evaluate the intensity of, and the impairment caused by pain. Four items measure pain intensity using 0 ("no pain") to 10 ("pain as bad as you can imagine") numeric rating scales, and 7 items measure the level of interference with function caused by pain using 0 (no interference) to 10 (complete interference) rating scales.
Adverse events assessments using NCI CTCAE (v5.0) | After first administration of study intervention up to 30 days after the last dose of study intervention
Incidence of fractures | Up to five years
Time to deterioration of FACT-P total score | Up to five years
  The FACT-P questionnaire assesses prostate cancer-related quality of life. The FACT-P total score is the sum of the scores of 39 items of the questionnaire and ranges from 1 to 156, the higher the score, the better the quality of life of prostate cancer patients.

CONTACTS AND LOCATIONS:
Locations (118):
- Australia (11):
  - Specialist Services Medical Group, Castle Hill, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - North West Cancer Centre, North Tamworth, New South Wales
  - Northern Cancer Institute, St Leonards, New South Wales
  - Prince of Wales Hospital NSW, Sydney, New South Wales
  - Illawarra Shoalhaven Local Health District, Wollongong, New South Wales
  - Icon Cancer Care, Brisbane, Queensland
  - Tasman Health Care, Southport, Queensland
  - The Tweed Hospital, Tugun, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
- Austria (2):
  - Klinik Ottakring - Wilhelminenspital, Vienna, Lower Austria
  - Kepler Universitätsklinikum Campus III, Linz, Upper Austria
- Czechia (7):
  - Fakultni nemocnice u sv. Anny, Brno
  - Krajska Zdravotní, a.s. - Nemocnice Chomutov, o.z. - Onkologické oddelení, Chomutov
  - Krajska Nemocnice Liberec, Liberec
  - Urocentrum Praha, s.r.o., Prague
  - Všeobecná fakultní nemocnice v Praze, Prague
  - Fakultni Thomayerova Nemocnice, Prague
  - Fakultní nemocnice Bulovka, Prague
- Finland (4):
  - OBSOLETE_Docrates Klinikka, Helsinki
  - Oulu University Hospital, Oulun yliopistollinen sairaala (OYS), Oulu
  - Seinäjoen keskussairaala, Seinäjoki
  - Tampere University Hospital, Tampereen yliopistollinen sairaala (TAYS), Tampere
- France (13):
  - Hôpital Saint André - Bordeaux, Bordeaux
  - Hôpital Morvan - Brest, Brest
  - Centre de Lutte Contre le Cancer François Baclesse, Caen
  - Hôpital Henri Mondor, Créteil
  - Centre Georges Francois Leclerc Dijon, Dijon
  - Centre Hospitalier Universitaire - Grenoble, Grenoble
  - Institut Paoli-Calmettes - Marseille, Marseille
  - Centre Antoine Lacassagne, Nice
  - Institut de Cancerologie Jean Godinot, Reims
  - Centre Eugène Marquis - Rennes Cedex, Rennes
  - CHU Strasbourg - Hopital Hautepierre, Strasbourg
  - Institut de Cancérologie de Lorraine - Alexis Vautrin, Vandœuvre-lès-Nancy
  - Gustave Roussy - Departement Oncologie-Radiotherapie, Villejuif
- Germany (2):
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate
- Hong Kong (5):
  - Pamela Youde Nethersole Eastern Hospital, Chai Wan, Hong Kong Island
  - Tuen Mun Hospital, Tuenmen, Hong Kong Island
  - Prince of Wales Hospital, Hong Kong, Hong Kong SAR
  - Queen Mary Hospital, Hong Kong, Hong Kong SAR
  - Hong Kong Integrated Oncology Centre (HKIOC), Central
- Hungary (2):
  - Semmelweis University, Budapest
  - Jasz-Nagykun-Szolnok Varmegyei Hetenyi Geza Korhaz, Szolnok
- Israel (2):
  - Lady Davis Carmel Medical Center, Haifa
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (10):
  - University Hospital Of Ferrara - Oncologia Clinica, Ferrara, Emilia-Romagna
  - Azienda Ospedaliero Universitaria di Modena_Policlinico - Oncologia, Modena, Emilia-Romagna
  - Azienda Ospedaliero Universitaria Parma - SC Oncologia Medica, Parma, Emilia-Romagna
  - Centro di Riferimento Oncologico di Aviano - Oncologia Medica e dei Tumori Immuno-Correlati, Aviano, Friuli Venezia Giulia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Servizio di Radioterapia Oncologica, Rome, Lazio
  - Ente Ospedaliero Ospedali Galliera Di Genova - Oncologia Medica, Genoa, Liguria
  - Istituto Europeo di Oncologia s.r.l, Milan, Lombardy
  - Azienda Ospedaliero-Universitaria Ss.Antonio E Biagio E C.Arrigo Alessandria_Presidio Civile - Oncologia, Alessandria, Piedmont
  - Azienda Provinciale Per I Servizi Sanitari_Ospedale Santa Chiara - UO Oncologia Medica, Trento, Trentino-Alto Adige
  - Istituto Oncologico Veneto_Padova - UOC Oncologia 1, Padua, Veneto
- Lithuania (4):
  - The Hospital of Lithuanian University of Health SciencesLUHS, Kaunas
  - PI Klaipedos University Hospital, Klaipėda
  - National Cancer Institute, Vilnius
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Poland (5):
  - Szpital Wojewodzki im. Mikolaja Kopernika w Koszalinie - Oddzial Dzienny Chemioterapii, Koszalin
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie, Krakow
  - Scanmed SA ZOZ Gastromed, Lublin
  - Szpital Grochowski im. dr.med. Rafala Masztaka, Warsaw
  - Uniwersytecki Szpital Kliniczny UM we Wroclawiu, Wroclaw
- Russia (2):
  - Chelyabinsk Regional Oncology Dispensary, Chelyabinsk
  - National Medical Research Radiology Center, Obninsk
- Singapore (2):
  - National Cancer Center Singapore - Oncology Department, Singapore
  - Singapore General Hospital, Singapore
- South Korea (5):
  - National Cancer Center, Goyang-si, Gyeonggido
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Seoul St. Mary's Hospital, Seoul, Seocho-Gu
  - Asan Medical Center | Ophthalmology, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
- Spain (16):
  - Complexo Hospitalario Universitario De Santiago | Oncologia, Santiago de Compostela, A Coruña
  - Hospital Universitari Son Espases | Oncologia, Palma de Mallorca, Balearic Islands
  - Hospital Germans Trias I Pujol | Oncologia, Badalona, Barcelona
  - Hospital General Universitario De Castellon | Oncologia, Castellon, Castellón
  - Hospital Universitario Puerta De Hierro De Majadahonda | Oncologia, Majadahonda, Madrid
  - Hospital Universitario Central De Asturias | Oncologia, Oviedo, Principality of Asturias
  - Fundacion Centro Oncologico Regional De Galicia Jose Antonio Quiroga Y Pineyro | Oncologia, A Coruña
  - Hospital Universitari Vall D Hebron | Oncologia, Barcelona
  - Institut Catala D'oncologia | Oncologia, Barcelona
  - Hospital De La Santa Creu I Sant Pau | Oncologia, Barcelona
  - Hospital Universitario Puerta Del Mar | Oncologia, Cadiz
  - Hospital Universitario De Jaen | Oncologia, Jaén
  - Hospital Universitario Lucus Augusti | Oncologia, Lugo
  - Hospital Universitario 12 De Octubre | Oncologia, Madrid
  - Hospital Universitario Virgen De La Victoria | Oncologia, Málaga
  - Fundacion Instituto Valenciano De Oncologia | Oncologia, Valencia
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital at Linkou, Taoyuan District
- Turkey (Türkiye) (19):
  - Baskent Universitesi Seyhan Hastanesi, Adana
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Ankara Yildirim Beyazit Universitesi Tip Fakültesi, Ankara
  - Ankara Universitesi Tip Fakultesi Hastanesi, Ankara
  - Trakya Univ. Tip Fak., Edirne
  - Gaziantep Universitesi Tip Fakultesi, Gaziantep
  - Istanbul Universitesi Istanbul Tip Fakultesi Hastanesi, Istanbul
  - Istanbul Egitim ve Arastirma Hastanesi, Istanbul
  - Istanbul Universitesi Cerrahpasa-Cerrahpasa Tip Fakultesi, Istanbul
  - TC Saglik Bakanligi Goztepe ProfDr Suleyman Yalcin Sehir Has, Istanbul
  - Medipol Universitesi Tip Fakultesi, Istanbul
  - Marmara University Medical Faculty | Pediatric Nephrology, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
  - Izmir Tepecik Egitim ve Arastirma Hastanesi, Izmir
  - Dokuz Eylul Universitesi Arastirma Uygulama Hastanesi, Izmir
  - Izmir Ekonomi Universitesi Medikal Point Hastanesi, Izmir
  - Erciyes Universitesi Tip Fakultesi, Kayseri
  - Mersin Universitesi Tip Fakultesi, Mersin
  - Ondokuz Mayis Universitesi Tip Fakultesi Saglik Uygulama ve Arastirma Merkezi, Samsun
- United Kingdom (2):
  - Royal Berkshire NHS Foundation Trust¦Royal Berkshire Hospital - Oncology, Reading, Berkshire
  - NHS Greater Glasgow & Clyde | Beatson West of Scotland Cancer Centre - Clinical Research Unit, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.